CLINICAL TRIAL: NCT01753310
Title: A Phase 3b, Multicentre, Randomised, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of DYSPORT® Using 2mL Dilution in Adults With Cervical Dystonia.
Brief Title: Efficacy and Safety of DYSPORT® Using 2mL Dilution in Adults With Cervical Dystonia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-TL-52120-169
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dysport® (Active Comparator): Dysport® (intramuscular injection), between 250 and 500 units (U)/vial using 2mL dilution, 1 cycle only
  Interventions: Biological: Botulinum toxin type A
- Placebo (Placebo Comparator): Placebo, up to 2mL
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — Intramuscular injection, between 250 and 500 units (U)/vial using 2mL dilution, 1 cycle only
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: Dysport®
Drug: Placebo — Up to 2mL
  Arms: Placebo

SUMMARY:
The purpose of the protocol is to evaluate the efficacy and safety of Dysport® using 2 mL dilution compared with placebo for the treatment of Cervical Dystonia.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Cervical Dystonia at least 9 months since onset and either previously untreated with botulinum toxin or currently treated with Botox at a total dosing range of 100-200 U and ≤60 U in the sternocleidomastoid muscle at the last injection cycle, and having had a satisfactory treatment response in the principal investigator's judgment during the last two sequential Botox treatment cycles.
* TWSTRS total score≥ 20; TWSTRS-severity subscale score> 10;

Exclusion Criteria:

* In apparent remission from Cervical Dystonia
* Diagnosis of pure retrocollis or pure anterocollis
* For non-naïve subjects, previous poor response to either of the last two Botox treatments
* Known requirement of <100U or >200U of Botox injected into the neck muscles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Neurology, M.D., Study Director — Ipsen
Locations (42):
- United States (42):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Movement Disorders Center of Arizona, LLC, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - East Bay Physician's Group, Berkeley, California
  - Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - Loma Linda University Healthcare, Department of Neurology, Loma Linda, California
  - USC Keck School of Medicine, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - University of Colorado at Denver Health Sciences, Aurora, Colorado
  - Advanced Neurosciences Research, Fort Collins, Colorado
  - Associated Neurologists of Southern Connecticut, Fairfield, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Parkinson's & Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Florida Center for Movement Disorders and Neurorestoration, Gainesville, Florida
  - Emerald Coast Center for Neurological Disorders, Pensacola, Florida
  - PD Treatment Center of SW FL, Port Charlotte, Florida
  - University of South Florida, Tampa, Florida
  - Guilford Neurologic Associates, West Palm Beach, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - NeuroTrials Research Inc., Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Kansas City Bone & Joint Clinic, Kansas City, Kansas
  - International Clinical Research Institute, Overland Park, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - Rehabilitation Consultants PA, Eagan, Minnesota
  - University of Medicine and Dentistry of New Jersey, Stratford, New Jersey
  - Atlantic Neuroscience Institute, Summit, New Jersey
  - Kingston Neurological Associates, Kingston, New York
  - Fazzini Parkinson's Disease & Dystonia Center, New York, New York
  - The Ichan School of Medicine at Mount Sinai, New York, New York
  - Island Neurological Associates, Plainview, New York
  - Guilford Neurologic Associates; Cone Health Medical Group, Greensboro, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - University of Cincinnati Physicians Company, LLC, Cincinnati, Ohio
  - OHSU Center for Health and Healing, Portland, Oregon
  - Penn State Hershey Neurology, Hershey, Pennsylvania
  - Coastal Neurology, Port Royal, South Carolina
  - North Texas Movement Disorders Institute, Bedford, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Puget Sound Neurology, Tacoma, Washington

REFERENCES:
- [Derived] Patel AT, Lew MF, Dashtipour K, Isaacson S, Hauser RA, Ondo W, Maisonobe P, Wietek S, Rubin B, Brashear A. Sustained functional benefits after a single set of injections with abobotulinumtoxinA using a 2-mL injection volume in adults with cervical dystonia: 12-week results from a randomized, double-blind, placebo-controlled phase 3b study. PLoS One. 2021 Feb 1;16(2):e0245827. doi: 10.1371/journal.pone.0245827. eCollection 2021. PMID 33524060

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 7 January 2013; last subject completed: 9 January 2015. 46 investigational sites in the United States of America were planned, 43 sites were initiated and 38 sites enrolled adult subjects with cervical dystonia (CD).
Pre-assignment Details: 150 subjects were screened; 16 subjects failed screening. 134 subjects were enrolled (signed informed consent) and were randomised with a 2:1 ratio of Dysport®:placebo. Randomisation was also stratified for subjects who were Botulinum toxin type A (BoNT-A) treatment naive or non-naive at baseline.
Groups:
- Dysport®: Subjects were randomised to receive a single intramuscular injected dose of study medication, Dysport® 500 U/vial using a 2 mL dilution scheme. The dose of Dysport® was between 250 U and 500 U divided among a minimum of two clinically indicated muscles. Dysport® contains the neurotoxin Clostridium botulinum type A toxin-hemagglutinin complex (abobotulinumtoxinA).
- Placebo: Subjects were randomised to receive a single dose of placebo by intramuscular injection. The placebo was provided in glass vials indistinguishable from the Dysport® vials. The placebo contained only the excipients used in Dysport® without the toxin, provided as a white lyophilised powder for reconstitution with the same storage and preparation conditions as for Dysport®.
Period: Overall Study
Arm/Group | Dysport® | Placebo
Started | 89 | 45
Completed | 57 | 21
Not Completed | 32 | 24
Not completed — Entered into open label extension study | 25 | 22
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Subject decision | 2 | 2
Not completed — Sponsor decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline characteristics are presented for the Intent to Treat (ITT) Population which consisted of all randomised subjects.
Arm/Group | Dysport® | Placebo | Total Title
Number analyzed (Participants) | 89 | 45 | 134
Age, Customized [Number; unit: participants]
  18-24 years | 0 | 0 | 0
  25-34 years | 2 | 2 | 4
  35-44 years | 9 | 4 | 13
  45-54 years | 26 | 14 | 40
  55-64 years | 26 | 12 | 38
  65-74 years | 22 | 11 | 33
  >75 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 28 | 87
  Male | 30 | 17 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Total Score at Week 4.
Description: The change from baseline in the TWSTRS total score at Week 4 was determined for the subjects who received a single dose of Dysport® or placebo by intramuscular injection at the baseline visit (Day 1), and is expressed as weighted overall treatment difference. The TWSTRS is an assessment scale used to measure the impact of CD on subjects, and comprises 3 subscales: severity, disability and pain, each of which is scored independently. The total score from the 3 subscales gives the TWSTRS total score with a value from 0 to 85 (best to worst). The score was assessed by the investigator prior to study treatment at baseline and at all post-treatment visits.
Time Frame: 4 weeks post-treatment
Population: The modified ITT population consisted of all randomised subjects with both a baseline and a Week 4 post-treatment TWSTRS total score assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport® | Placebo
Number analyzed (Participants) | 84 | 45
units on a scale
  Baseline (Day 1) Pre-treatment | 42.5 (10.40) | 42.4 (10.63)
  Week 4 Post-treatment | 31.7 (15.29) | 39.9 (12.46)
Statistical Analysis 1: Comparison: Dysport® vs Placebo; The superiority of Dysport® to placebo was tested at a two-tailed 5% level by using a stratified analysis of covariance (ANCOVA) with baseline TWSTRS total score as covariate and stratified by the randomisation stratification factor (BoNT-A naïve versus BoNT-A non-naïve); Test type: Superiority or Other; p < 0.001, t-test, 2 sided; The 2 sided t-test was on weighted overall treatment difference; Mean Difference = -8.3, 95% CI 2-sided [-12.17 to -4.47], Standard Error of Mean 1.95 — Based on the sample size weighted overall treatment difference

2. Secondary Outcome: Change From Baseline in TWSTRS Total Score at Week 2.
Description: The change from baseline in the TWSTRS total score at Week 2 was determined for the subjects who received a single dose of Dysport® or placebo by intramuscular injection at the baseline visit (Day 1), and is expressed as weighted overall treatment difference. The TWSTRS is an assessment scale used to measure the impact of CD on subjects, and comprises 3 subscales: severity, disability and pain, each of which is scored independently. The total score from the 3 subscales gives the TWSTRS total score with a value from 0 to 85 (best to worst). The score was assessed by the investigator prior to study treatment at baseline and at all post-treatment visits.
Time Frame: 2 weeks post-treatment
Population: The ITT population consisted of all randomised subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport® | Placebo
Number analyzed (Participants) | 89 | 45
units on a scale
  Baseline (Day 1) pre-treatment | 42.1 (10.77) | 42.4 (10.63)
  Week 2 post-treatment | 34.5 (14.54) | 39.8 (12.72)
Statistical Analysis 1: Comparison: Dysport® vs Placebo; The superiority of Dysport® to placebo was tested at a two-tailed 5% level by using a stratified ANCOVA with baseline TWSTRS total score as covariate and stratified by the randomisation stratification factor (BoNT-A naïve versus BoNT-A non-naïve); Test type: Superiority or Other; p = 0.001, t-test, 2 sided; The 2 sided t-test was on weighted overall treatment difference; Mean Difference = -5.4, 95% CI 2-sided [-8.67 to -2.14], Standard Error of Mean 1.65 — Based on the sample size weighted overall treatment difference

3. Secondary Outcome: Change From Baseline in Clinical Global Impression of Change (CGIC) in CD at Week 2.
Description: The CGIC is an investigator-reported assessment of the global clinical change in CD since study treatment administration. The CGIC uses a seven-point Likert scale ranging from +3 (very much improved) to -3 (very much worse), and was assessed by the investigator at the Week 2 and Week 4 visits.
Time Frame: 2 weeks post-treatment
Population: The ITT population consisted of all randomised subjects. Only subjects with data available at the point of testing are reported. A total of 4 subjects (3 from the Dysport® arm and 1 from the Placebo arm) had missing values for CGIC.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport® | Placebo
Number analyzed (Participants) | 86 | 44
units on a scale | 1.2 (1.32) | -0.0 (1.07)
Statistical Analysis 1: Comparison: Dysport® vs Placebo; The superiority of Dysport® to placebo on CGIC of CD was tested at a two-tailed 5% level by using an analysis of variance (ANOVA) with treatment and randomisation stratification factor as main effects; Test type: Superiority or Other; p < 0.001, ANOVA

4. Secondary Outcome: TWSTRS Responders at Week 2.
Description: Treatment response was determined as the number of responders at Week 2 relative to the baseline TWSTRS total score. A treatment responder is defined as a subject who had at least a 30% reduction in the TWSTRS total score after treatment. This was calculated as ([Week 2 score - baseline score]/baseline score) * 100.
Time Frame: 2 weeks post-treatment
Population: The ITT population consisted of all randomised subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dysport® | Placebo
Number analyzed (Participants) | 89 | 45
percentage of participants | 27.9 [18.8 to 38.6] | 11.4 [3.8 to 24.6]
Statistical Analysis 1: Comparison: Dysport® vs Placebo; The superiorty of Dysport® to placebo on treatment response was tested at a two-tailed 5% level by using a Mantel-Haenszel chi-squared test stratified by the randomisation factor; Test type: Superiority or Other; p = 0.033, Mantel-Haenszel chi-squared test

5. Secondary Outcome: Change From Baseline in CGIC in CD at Week 4.
Description: as for outcome 3
Time Frame: 4 weeks post-treatment
Population: The ITT population consisted of all randomised subjects. Only subjects with data available at the point of testing are reported. A total of 3 subjects (all from the Dysport® arm) had missing values for CGIC.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport® | Placebo
Number analyzed (Participants) | 86 | 45
units on a scale | 1.2 (1.50) | 0.1 (1.27)
Statistical Analysis 1: Comparison: Dysport® vs Placebo; The superiority of Dysport® to placebo on CGIC of CD was tested at a two-tailed 5% level by using an ANOVA with treatment and randomisation stratification factor as main effects; Test type: Superiority or Other; p < 0.001, ANOVA

6. Secondary Outcome: TWSTRS Responders at Week 4.
Description: Treatment response was determined as the number of responders at Week 4 relative to the baseline TWSTRS total score. A treatment responder is defined as a subject who had at least a 30% reduction in the TWSTRS total score after treatment. This was calculated as ([Week 4 score - baseline score]/baseline score) * 100.
Time Frame: 4 weeks post-treatment
Population: The ITT population consisted of all randomised subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dysport® | Placebo
Number analyzed (Participants) | 89 | 45
percentage of participants | 41.9 [31.3 to 53.0] | 11.1 [3.7 to 24.1]
Statistical Analysis 1: Comparison: Dysport® vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mantel-Haenszel chi-squared test

7. Secondary Outcome: Change From Baseline in Cervical Dystonia Impact Profile-58 (CDIP-58) Total Score at Week 4.
Description: The CDIP-58 scale is a subject-based rating scale measuring the health impact of CD measured in 8 health dimensions including head and neck symptoms, pain and discomfort, upper limb activities, walking, sleep, annoyance, mood and psychosocial functioning. Subscale scores were transformed to a common theoretical range of 0 (no impact) to 100 (most impact). Negative changes from the baseline total score indicate improvement in the impact of CD on health whereas postive changes indicate worsening.
Time Frame: 4 weeks post-treatment
Population: The ITT population consisted of all randomised subjects. Only subjects with data available at the point of testing are reported. A total of 8 subjects (7 from the Dysport® arm and 1 from the Placebo arm) had missing values for CDIP-58.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport® | Placebo
Number analyzed (Participants) | 82 | 44
units on a scale | -8.5 (14.26) | -4.7 (16.18)
Statistical Analysis 1: Comparison: Dysport® vs Placebo; The superiority of Dysport® to placebo on CDIP-58 was tested at a two-tailed 5% level by using an ANOVA with treatment and randomisation stratification factor as main effects; Test type: Superiority or Other; p = 0.174, ANOVA

8. Secondary Outcome: Change From Baseline in CDIP-58 Total Score at Week 2.
Description: The CDIP-58 scale is a subject-based rating scale measuring the health impact of CD measured in 8 health dimensions including head and neck symptoms, pain and discomfort, upper limb activities, walking, sleep, annoyance, mood and psychosocial functioning. Subscale scores were transformed to a common theoretical range of 0 (no impact) to 100 (most impact). Negative changes from the baseline total score indicate improvement in the impact of CD on health whereas postive changes indicate worsening. The hierarchical testing procedure would only be conducted if the previous secondary efficacy endpoint (change from baseline in CDIP-58 total score at Week 4) reached a statistically significant treatment effect. This secondary efficacy endpoint (change from baseline in CDIP-58 total score at Week 2) was performed to characterise the full clinical effect.
Time Frame: 2 weeks post-treatment
Population: The ITT population consisted of all randomised subjects. Only subjects with data available at the point of testing are reported. A total of 8 subjects (6 from the Dysport® arm and 2 from the Placebo arm) had missing values for CDIP-58.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport® | Placebo
Number analyzed (Participants) | 83 | 43
units on a scale | -5.8 (13.96) | -4.3 (14.49)
Statistical Analysis 1: Comparison: Dysport® vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.583, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of informed consent to end of study/early withdrawal (period of up to 13 weeks).
Description: Serious and non-serious treatment emergent AEs (TEAEs) are presented. The safety population consisted of all randomised subjects who received study treatment regardless of the amount of study treatment administered and who had at least one follow up safety assessment.
Arm/Group | Dysport® | Placebo
Serious Adverse Events (participants affected / at risk) | 4/88 | 1/45
Other Adverse Events (participants affected / at risk) | 35/88 | 10/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport® (N=88) | Placebo (N=45)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport® (N=88) | Placebo (N=45)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8 (8) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 7 (7) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Burning sensation (Nervous system disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 2 (2)
Post injection phenomenon (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No